CLINICAL TRIAL: NCT04024709
Title: Long-term Results of Per-oral Pyloromyotomy for Refractory Gastroparesis
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_0033
Record Dates: First submitted 2019-07-09; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Gastroparesis
Keywords: G-POEM; gastroparesis; POP; oral endoscopic pyloromyotomy
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Gastric Peroral Endoscopic Myotomy — Creation by submucosal dissection of a tunnel in the gastric wall at the level of the antrum, then of a pyloric and antral myotomy, before closing the mucosal access by clips.

SUMMARY:
This is a large multicenter retrospective French cohort conducted in seven French centers that had performed at least five G-POEM procedures at the end of 2017. All patients treated by G-POEM for refractory gastroparesis since April 30, 2014 (first case of GPOEM in France) in these seven centers were included in this study and followed until April 2019. The data were collected retrospectively regarding medical and technical data, and then prospectively for the following data, which were included in a database for each center and combined for analysis.

Gastric Cardinal Symptoms Index (GCSI) was used to evaluate symptoms and their severity. It applies a Likert scale ranging from 0 to 5 (5 being the highest score) for three subscales: satiety (mean of four items), nausea/vomiting (mean of three items), and bloating (mean of two items). The total GCSI score was the mean of the three subscales. A GCSI score ≥ 2.6 is considered moderate gastroparesis and ≥ 3 is considered severe.

Gastric emptying scintigraphy (GES) was used to confirm delayed gastric emptying, since it is considered the gold standard according to the American Society of Neurogastroenterology. Patients consume a radiolabeled meal, receive imaging at specific time-points to determine gastric retention. The exam is pathological when retention is > 90% after 1 hour, > 60% after 2 hours (H2), > 30% after 3 hours (H3), and > 10% after 4 hours (H4). All but one center performed the GES according to the US guidelines: that center performed a 3-hour GES with a local validation of a threshold of 30% retention at H3 to define delayed gastric emptying. A %H4 retention > 30% was defined as severe delayed gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* treatment by G-POEM during the study period,
* at least a 1-year follow-up, and
* GCSI evaluation before and 1 year after G-POEM.

Exclusion Criteria:

* missing GCSI before and/or 12 months after G-POEM,
* non-pathological GES before G-POEM: delayed gastric emptying was defined as t ½ > 113 min and %H4 retention > 10%, and
* loss to follow-up or death before 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastroparesis
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical success of G-POEM | 1 year
  evaluate the clinical success at the 1-year follow-up, defined by a decrease in the GCSI score by at least 1 point compared to baseline.

SECONDARY OUTCOMES:
Incidence of adverse events of pylorotomy | 2 years
  analysis of adverse events during the two years following the pylorotomy (including perforation per-gesture, bleeding post-gesture). ASGE lexicon will be used to grade these adverse events
Clinical success of G-POEM | 2 years
  evaluate the clinical success at the 1-year follow-up, defined by a decrease in the Gastroparesis Cardinal Symptoms Index score by at least 1 point compared to baseline. GCSI is a Likert scale ranging from 0 to 5 (5 being the worst score) for three subscales: satiety (mean of four items), nausea/vomiting (mean of three items), and bloating (mean of two items). The total GCSI score was the mean of the three subscales. A GCSI score ≥ 2.6 is considered moderate gastroparesis and ≥ 3 is considered severe.
Delayed gastric emptying after the procedure | 2 years
  Gastric emptying scintigraphy (GES) was used to confirm delayed gastric emptying, since it is considered the gold standard according to the American Society of Neurogastroenterology. Patients consume a radiolabeled meal, receive imaging at specific time-points to determine gastric retention. The exam is pathological when retention is > 90% after 1 hour, > 60% after 2 hours (H2), > 30% after 3 hours (H3), and > 10% after 4 hours (H4). Percent retention at 2hours and 4hours will be compared before and after the procedure.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - University Hospital, Lille
  - University Hospital, Limoges
  - Hospices Civiles Lyon, Lyon
  - University Hospital, Marseille
  - University Hospital, Nice
  - Cochin Hospital, Paris
  - University Hospital, Rennes

REFERENCES:
- [Background] Gonzalez JM, Benezech A, Vitton V, Barthet M. G-POEM with antro-pyloromyotomy for the treatment of refractory gastroparesis: mid-term follow-up and factors predicting outcome. Aliment Pharmacol Ther. 2017 Aug;46(3):364-370. doi: 10.1111/apt.14132. Epub 2017 May 15. PMID 28504312
- [Background] Khashab MA, Ngamruengphong S, Carr-Locke D, Bapaye A, Benias PC, Serouya S, Dorwat S, Chaves DM, Artifon E, de Moura EG, Kumbhari V, Chavez YH, Bukhari M, Hajiyeva G, Ismail A, Chen YI, Chung H. Gastric per-oral endoscopic myotomy for refractory gastroparesis: results from the first multicenter study on endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2017 Jan;85(1):123-128. doi: 10.1016/j.gie.2016.06.048. Epub 2016 Jun 25. PMID 27354102
- [Background] Jacques J, Pagnon L, Hure F, Legros R, Crepin S, Fauchais AL, Palat S, Ducrotte P, Marin B, Fontaine S, Boubaddi NE, Clement MP, Sautereau D, Loustaud-Ratti V, Gourcerol G, Monteil J. Peroral endoscopic pyloromyotomy is efficacious and safe for refractory gastroparesis: prospective trial with assessment of pyloric function. Endoscopy. 2019 Jan;51(1):40-49. doi: 10.1055/a-0628-6639. Epub 2018 Jun 12. PMID 29895073
- [Background] Revicki DA, Camilleri M, Kuo B, Szarka LA, McCormack J, Parkman HP. Evaluating symptom outcomes in gastroparesis clinical trials: validity and responsiveness of the Gastroparesis Cardinal Symptom Index-Daily Diary (GCSI-DD). Neurogastroenterol Motil. 2012 May;24(5):456-63, e215-6. doi: 10.1111/j.1365-2982.2012.01879.x. Epub 2012 Jan 27. PMID 22284754
- [Background] Abell TL, Camilleri M, Donohoe K, Hasler WL, Lin HC, Maurer AH, McCallum RW, Nowak T, Nusynowitz ML, Parkman HP, Shreve P, Szarka LA, Snape WJ Jr, Ziessman HA; American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. Consensus recommendations for gastric emptying scintigraphy: a joint report of the American Neurogastroenterology and Motility Society and the Society of Nuclear Medicine. J Nucl Med Technol. 2008 Mar;36(1):44-54. doi: 10.2967/jnmt.107.048116. Epub 2008 Feb 20. PMID 18287197
- [Background] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521
- [Derived] Ragi O, Jacques J, Branche J, Leblanc S, Vanbiervliet G, Legros R, Pioche M, Rivory J, Chaussade S, Barret M, Wallenhorst T, Barthet M, Kerever S, Gonzalez JM. One-year results of gastric peroral endoscopic myotomy for refractory gastroparesis: a French multicenter study. Endoscopy. 2021 May;53(5):480-490. doi: 10.1055/a-1205-5686. Epub 2020 Jul 21. PMID 32575130